CLINICAL TRIAL: NCT04563195
Title: BAFF/IL-17 Bispecific Antibody Treatment in Subjects With Primary Sjogren's Syndrome
Acronym: BAFF/IL-17
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Drug unavailable
Sponsor: Matthew C. Baker (Other)
Responsible Party: Sponsor-Investigator, Matthew C. Baker, Clinical Assistant Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 56505
Record Dates: First submitted 2020-09-12; First posted 2020-09-24 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Primary Sjogren's Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- open label (Other): open label study; all subjects will receive the same drug at the same dose
  Interventions: Drug: tibulizumab (LY3090106)

INTERVENTIONS:
Drug: tibulizumab (LY3090106) — subcutaneous injections of 300mg every 2 weeks over a period of 12 weeks
  Other Names: open label

SUMMARY:
To demonstrate that tibulizumab (LY3090106) treatment improves the mean unstimulated salivary flow rate or the salivary gland total ultrasound score (TUS) in primary Sjogren's syndrome patients at week 12 compared to the baseline visit.

DETAILED DESCRIPTION:
This will be a single-site, open-label study in patients with primary Sjogren's syndrome. All patients will receive tibulizumab (LY3090106) 300mg subcutaneously every 2 weeks for a total of 12 weeks.

Primary Sjogren's syndrome was selected as a relevant patient population based on the mechanism of action of the molecule and the current understanding of the pathogenesis of the disease. An open-label design was chosen based on practical considerations regarding the number of patients that could be recruited. Although open-label studies are subject to bias, objective primary endpoints were intentionally chosen to minimize this concern.

The goal of this study is to demonstrate that tibulizumab (LY3090106) treatment improves the mean unstimulated salivary flow rate or the salivary gland total ultrasound score (TUS) in primary Sjogren's syndrome patients at week 12 compared to the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-85 years of age
* Confirmed diagnosis of primary Sjogren's syndrome by the 2016 ACR-EULAR classification criteria for primary Sjogren's syndrome
* All women (regardless of childbearing potential) must test negative for pregnancy at the time of screening
* Women must also agree to use a reliable method of birth control from screening until 12 weeks following last dose of study drug unless they are not of child bearing potential
* Have stimulated whole salivary flow rate of greater than or equal to 0.10 ml/minute
* Have a salivary gland total ultrasound score (TUS) of less than or equal to 9 (on a 0-11 point scale)

Exclusion Criteria:

* Currently enrolled in a clinical trial involving an investigational product or off-label use of a drug
* Concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have received any nonbiologic investigational product within 30 days or 5 half-lives (whichever is longer) of their baseline (Day 1) visit
* Have received any biologic investigational product within 3 months or 5 half-lives (whichever is longer) of their baseline visit, or any leukocyte depleting agent within 12 months of baseline
* Have disease-modifying antirheumatic drug (DMARD) or immunosuppressive use as follows:

  * ANY treatment with a janus kinase (JAK) inhibitor (including but not limited to tofacitinib, baricitinib, upadacitinib, or filgotinib) within 28 days prior to baseline or planned treatment with a JAK inhibitor during the study
  * UNSTABLE PRESCRIBED DOSE of other synthetic DMARDs (eg, hydroxychloroquine, methotrexate, leflunomide, or sulfasalazine) within 28 days prior to baseline or if the dose of drug is planned to be increased during the study (stable prescriptions are allowed)
  * ANY treatment with cytotoxic or immunosuppressive drugs including but not limited to cyclophosphamide, mycophenolic acid, azathioprine, cyclosporine, sirolimus, or tacrolimus within 28 days prior to screening or planned treatment during the study
  * Have had treatment with biologic DMARDs as follows: Etanercept, adalimumab, or anakinra <4 weeks before baseline or planned treatment during the study
  * Have had treatment with biologic DMARDs as follows: Infliximab, certolizumab pegol, golimumab, abatacept, or tocilizumab <8 weeks before baseline or planned treatment during the study
* Are persons who have previously completed or withdrawn from this study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
whole unstimulated sialometry | baseline
  change in unstimulated salivary flow
whole unstimulated sialometry | week 12
  change in unstimulated salivary flow
salivary gland ultrasound | baseline
  change in salivary gland ultrasound score
salivary gland ultrasound | week 12
  change in salivary gland ultrasound score

SECONDARY OUTCOMES:
ESSDAI | baseline
  change in the ESSDAI disease activity score
  The EULAR Sjogren's Syndrome Disease Activity Index (ESSDAI) is a physician administered questionnaire containing 12 organ-specific domains designed to measure disease activity. The ESSDAI score is obtained by addition of the twelve domain scores. Each domain score is obtained by multiplying the activity level with the domain weight. The maximum theoretical ESSDAI score is 123 and the minimum score is 0. A higher score means more disease activity (worse outcome).
ESSDAI | week 12
  change in the ESSDAI disease activity score
  The EULAR Sjogren's Syndrome Disease Activity Index (ESSDAI) is a physician administered questionnaire containing 12 organ-specific domains designed to measure disease activity. The ESSDAI score is obtained by addition of the twelve domain scores. Each domain score is obtained by multiplying the activity level with the domain weight. The maximum theoretical ESSDAI score is 123 and the minimum score is 0. A higher score means more disease activity (worse outcome).
ESSPRI | baseline
  change in the ESSPRI disease activity score
  The EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI) is a patient completed questionnaire to assess subjective patient symptoms, which includes 3 domains (dryness, fatigue, and pain). The ESSPRI score is calculated by averaging the three domains with a maximum severity score of 10 and minimum score of 0. A higher score means more disease activity (worse outcome).
ESSPRI | week 12
  change in the ESSPRI disease activity score
  The EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI) is a patient completed questionnaire to assess subjective patient symptoms, which includes 3 domains (dryness, fatigue, and pain). The ESSPRI score is calculated by averaging the three domains with a maximum severity score of 10 and minimum score of 0. A higher score means more disease activity (worse outcome).
whole stimulated sialometry | baseline
  change in stimulated salivary flow rate
whole stimulated sialometry | week 12
  change in stimulated salivary flow rate
Schirmer I test | baseline
  change in the Schirmer I test
Schirmer I test | week 12
  change in the Schirmer I test
MRI | baseline
  change in MRI (parenchymal architecture scored 0 to 4 and sialography scored 0 to 4)
MRI | week 12
  change in MRI (parenchymal architecture scored 0 to 4 and sialography scored 0 to 4)
PET | baseline
  change in PET (parotid and submandibular gland SUVmax)
PET | week 12
  change in PET (parotid and submandibular gland SUVmax)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No